CLINICAL TRIAL: NCT00015626
Title: A Clinical Trial to Prevent the Complications of Insulin Resistance (Including Type-2 Diabetes)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NCRR-M01RR06020-0057
Record Dates: First submitted 2001-04-24; First posted 2001-04-26 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Insulin Resistance; Diabetes Mellitus
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus | interventions — Metformin; Diet; Exercise; Pioglitazone; Rosiglitazone

INTERVENTIONS:
Drug: Metformin
Procedure: skin biopsy
Behavioral: diet and exercise
Drug: pioglitazone
Drug: rosiglitazone

SUMMARY:
The goal of this study is to aggressively treat insulin resistance and its clinical manifestations when they first appear in childhood, and to prevent the subsequent progression towards impaired glucose tolerance and type-2 diabetes. In the process of this clinical trial, we will learn more about the early manifestations of insulin resistance, its treatment, and its relationship to obesity and type-2 diabetes through parallel in-vivo and in-vitro studies.

ELIGIBILITY:
Inclusion criteria:

1. Obese patients (wt > 95th percentile for age, for adults increased BMI > 27) greater than 5 years of age
2. And/or presence of complications of insulin resistance such as acanthosis nigricans, dyslipidemia, elevated blood pressure, hyperandrogenism
3. Siblings and parents of patients with insulin resistance. Siblings and parents will be included only in the case of documented insulin resistance in the index subject. Insulin resistance will be documented by OGTT and/or IVGTT.
4. Family history of type II diabetes.

Exclusion Criteria:

1. Critically ill patients, patients will congestive heart failure, renal or liver insufficiency
2. Inability to give consent.
3. History of poor compliance with physician's recommendations

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300

CONTACTS AND LOCATIONS:
Locations (1):
- Cornell University, New York, New York, United States

REFERENCES:
- [Derived] Ipsen EO, Madsen KS, Chi Y, Pedersen-Bjergaard U, Richter B, Metzendorf MI, Hemmingsen B. Pioglitazone for prevention or delay of type 2 diabetes mellitus and its associated complications in people at risk for the development of type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 19;11(11):CD013516. doi: 10.1002/14651858.CD013516.pub2. PMID 33210751